CLINICAL TRIAL: NCT03928626
Title: Brief ROC Training Effects on Alcohol Drinking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to COVID shutting down all research at Yale University.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000023367
Record Dates: First submitted 2019-04-11; First posted 2019-04-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Binge Drinking; Heavy Drinking; Young Adult; Heavy Drinker; Alcohol Drinking; Alcohol Drinking in College; Drinking Behavior; Drunkenness; Drinking Excessive; Drinking Problem; Drink Too Much; College Drinking
Keywords: Binge Drinking; Heavy Drinking; Young Adult; Heavy Drinker; Regulation of craving; Cognitive behavioral therapy; Neurocognitive training; Emotion regulation; Alcohol
MeSH Terms: conditions — Binge Drinking; Alcoholic Intoxication; Alcohol Drinking; Alcohol Drinking in College; Drinking Behavior; Alcoholism; Emotional Regulation | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRAVING REGULATION (Active Comparator): In the CRAVING REGULATION condition, participants will first read a brief essay about the adverse consequences of drinking alcohol. Then, participants may complete a comprehension check consisting of questions to ensure that they understood and encoded the content of the essays. Participants will be trained to use the information to inform the strategy they will use in the regulation of craving training (ROC-T). A single trial in the regulation of craving training will have two possible instructions: (a) STRATEGY: implement the strategy ("bring to mind the negative facts from the essay") and (b) LOOK: to merely observe the image and allow natural responses to come. Participants will follow the instructions; followed by an alcohol-related picture, a brief delay, and will then rate their craving. Participants will then be instructed to use this strategy in daily life situations when they might drink.
  Interventions: Behavioral: Regulation of craving
- CONTROL (NO REGULATION) (Placebo Comparator): In the CONTROL condition, participants will first read a brief essay about a non-alcohol-related topic (e.g., color perception). Then, participants will complete a comprehension check consisting of questions to ensure that they understood and encoded the content of the essays. Participants will view images of objects that are unrelated to alcohol. Furthermore, participants in the control condition will not practice any strategy in the regulation of craving task (ROC-T). That is, in the CONTROL condition, participants would merely observe the image and allow natural responses to come (i.e., LOOK instruction) and rate how colorful is each item (this controls for task time and experiment setting).
  Interventions: Behavioral: Control (NO REGULATION)

INTERVENTIONS:
Behavioral: Regulation of craving — Participants in the ROC-T condition will be trained to use a strategy that instructs them to think of the negative outcomes associated with alcohol drinking while looking at alcohol-related images.
  Other Names: Neurocognitive training
  Arms: CRAVING REGULATION
Behavioral: Control (NO REGULATION) — In the CONTROL condition, participants would simply observe non-alcohol-related images and allow natural responses to come
  Other Names: Sham (No regulation)
  Arms: CONTROL (NO REGULATION)

SUMMARY:
The goal of the proposed study is to examine whether a single session of training in regulation of craving (ROC-T) affects alcohol drinking. The study will consist of (1) a basic screening (phone and/or online) and an in-person visit, to determine eligibility and conduct pre-intervention baseline assessments; (2) a training (ROC-T) visit, (3) a post-intervention assessment visit, and (4) 1-2 phone/online follow-up assessments.

The study will take up to 10 hours of the participants' time.

DETAILED DESCRIPTION:
The investigators propose to test the efficacy of such training by randomizing 120 individuals who report alcohol drinking to the following conditions: (1) a brief training in cognitive regulation and (2) a control or no-training condition. Training will be delivered in a computerized session (approximately 60 minutes). If randomized into the cognitive regulation training, subjects will be trained to use a cognitive strategy while viewing images of alcoholic drinks. The strategy would be to follow instructions to think about the adverse outcomes associated with continued alcohol drinking. If randomized into the control condition, participants will only view non-alcohol-related images with no use of strategy. After all the training sessions are completed, participants will complete several follow-ups. The investigators will evaluate the effects of training on alcohol drinking pre- and post-training.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-25
2. Capability of performing the experimental tasks (e.g., can read, able to use computers)
3. Native or fluent speaker of English
4. Provides informed consent
5. Normal or corrected-to-normal vision
6. Willing to commit to the full length of the protocol
7. Heavy drinking or binge-drinking

Exclusion Criteria.

1. Present DSM disorders, apart from alcohol use disorders
2. Reports of neurological or systemic disorders that can cause cognitive impairment
3. Minor cognitive impairment evidenced by an inability to correctly understand study information
4. Reports entirely no interest in reducing the amount of drinking (Alcohol Contemplation Ladder score of 9 or 10).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Timeline followback (TLFB) | Baseline (first visit) to post-intervention (an average of one week after first visit)
  The Alcohol TLFB is a drinking assessment method that obtains estimates of daily drinking.

SECONDARY OUTCOMES:
Frequency of regulating drinking + craving. | Will be measured at post-intervention (one week after first visit)
  Participants will be asked to report their craving regulation (if any) since the intervention. In order to assess the level of craving regulation the participants will answer several questions in our craving regulation questionnaire. This assessment will include questions about the number of attempts at craving regulation, the number of times the participant intended to regulate craving, one's confidence in one's ability to regulate craving, the level of motivation to regulate drinking before each drinking episode, and the participant's intention to regulate drinking in the future. Finally, participants will be asked how many times they were thinking of negative consequences in general and while experiencing alcohol craving.
Timeline followback (TLFB) | First visit, post-intervention (one week after first visit), follow-up (two weeks after first visit)
  The Alcohol TLFB is a drinking assessment method that obtains estimates of daily drinking.

CONTACTS AND LOCATIONS:
Overall Officials: Uri Berger, PhD, Study Director — Yale University
Locations (1):
- Clinical & Affective Neuroscience Lab, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.